CLINICAL TRIAL: NCT07277803
Title: Effects of Device-Based and Manual Sensory Acuity Training on Chronic Low Back Pain: A Three-Arm Randomized Controlled Trial Protocol
Brief Title: Device-Based vs Manual Sensory Training in Low Back Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, AYŞE GÜRLÜK, PhD Student, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MedipolUniversity2025; 225S070 (Other Grant/Funding Number: TUBITAK)
Record Dates: First submitted 2025-05-27; First posted 2025-12-11 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Low Back Pain
Keywords: Chronic pain; physiotherapy and rehabilitation; radial/local vibration; low back pain; pain treatment; tactile feedback; mobile applications; wearable technologies; embedded system design
MeSH Terms: conditions — Low Back Pain; Chronic Pain; Agnosia | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: This is an interventional randomized controlled trial with parallel assignment. The study was designed as a single-blind study; only the clinical evaluator will be blinded. Participants and therapists administering the intervention will not be blinded due to the nature of the intervention. The evaluator's lack of knowledge about group assignments was planned to ensure objectivity of the measurements and minimize the risk of bias. Patients and the public were not involved in the design or conduct of this trial. The study design and intervention protocols were informed by existing scientific evidence and clinical guidelines. Participant burden was considered in determining session duration and assessment procedures. Participants will not be involved in the interpretation or dissemination of the study findings.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes

ARMS (3):
- Manual Sensory Acuity Training Group (M-SATG) (Experimental): In addition to motor control exercises, individuals with NLBP included in the M-SATG will receive sensory acuity training with progressively increasing levels of difficulty. This training will include manually administered components of localization acuity, orientation acuity, temporal acuity, and graphesthesia. All sensory acuity components (localization, orientation, temporal acuity, graphesthesia) will be delivered in randomized sequences generated prior to each session. During localization, orientation, and temporal acuity tasks, a standardized adhesive grid template consisting of 16 points will be applied to the lumbar region to guide stimulus delivery. Throughout the training process, participants will progress to the next training stage once they achieve 80% accuracy for that week. A response interval of 10 seconds will be provided between stimuli, with 1 minute rest periods between training sets and 2 minute rest periods between different training parameters.
  Interventions: Other: Manual Sensory Acuity Training Group (M-SATG)
- Control Group (CG) (Experimental): All individuals in this group will receive Motor Control Exercises (MCEs) for 30 minutes to promote correct muscle activation, postural alignment, movement integrity, and optimal control of the spine and pelvis. In addition to MCEs, participants will also receive a structured 30-minute patient education (PE) program, matched to the duration of the structured SAT program administered in the other groups. The PE program will focus on developing safe movement strategies, postural awareness, ergonomics, and self-management skills.
  Interventions: Other: Control Group (CG)
- Technology-Based Sensory Acuity Training Group (T-SATG) (Experimental): Participants in this arm will receive technology-based sensory acuity training delivered through the TactiPain device in addition to motor control exercises. The training will include vibrotactile localization, orientation, temporal acuity, and graphesthesia tasks administered with a progressive weekly protocol. Vibrotactile stimuli will be presented through a 4×4 matrix of 16 vibration motors positioned over the lumbar region, with weekly progression in intensity, vibration duration, and inter-stimulus intervals. Randomized sequences will be used for all tasks, and progression will occur when ≥80% accuracy is achieved. A response interval of 10 seconds will be provided between stimuli, with 1 minute rest periods between training sets and 2 minute rest periods between different training parameters.
  Interventions: Device: Technology-Based Sensory Acuity Training Group (T-SATG)

INTERVENTIONS:
Device: Technology-Based Sensory Acuity Training Group (T-SATG) — The vibrotactile stimuli will be delivered according to a predefined weekly progression. In Week 1, high-intensity vibrations will be applied with a duration of 500 ms and an inter-stimulus interval of 1 second. In Week 2, medium-intensity vibrations will be delivered with a duration of 500 ms and a 500-ms inter-stimulus interval. In Week 3, medium-intensity vibrations will be delivered with a duration of 200 ms and a 200-ms inter-stimulus interval, and in Week 4, low-intensity vibrations will be applied with a duration of 100 ms and a 100-ms inter-stimulus interval. This structured progression is designed to ensure a gradual increase in task difficulty and to standardize the vibrotactile training across participants.
  Arms: Technology-Based Sensory Acuity Training Group (T-SATG)
Other: Control Group (CG) — The MCE program will follow a progressive approach targeting activation of the transversus abdominis and multifidus muscles. It will begin with basic exercises emphasizing isolated contractions and progress to more complex movements involving co-activation of both muscles, including bridging and quadruped exercises. As part of the PE component, participants will receive fundamental information regarding spinal health, neutral spine posture, and appropriate movement strategies for daily activities. Guidance will be provided on ergonomics, including lifting techniques, workspace organization, and methods to reduce mechanical load on the lower back. The program will also support self-care by promoting regular physical activity, appropriate pacing during flare-ups, adequate rest, and healthy lifestyle habits.
  Arms: Control Group (CG)
Other: Manual Sensory Acuity Training Group (M-SATG) — To progressively increase difficulty, Semmes-Weinstein monofilaments with thick and thin tips will be used to vary stimulus pressure. Stimulus duration will advance weekly: week 1 - thick tip 5 s, week 2 - thick tip 2 s, week 3 - thin tip 5 s, week 4 - thin tip 2 s, with a stopwatch ensuring standardization and fixed intervals between stimuli. All sensory acuity tasks (localization, orientation, temporal acuity, and graphesthesia) will be delivered using randomized sets generated by random.org to prevent habituation. Responses will be recorded weekly to track progress. An adhesive 16-hole grid template will be placed between the last rib and sacrum on each participant before each session.
  Arms: Manual Sensory Acuity Training Group (M-SATG)

SUMMARY:
Chronic low back pain (CLBP) is a leading cause of disability worldwide and affects a large proportion of working-age individuals. Cortical reorganization in CLBP, particularly within the sensorimotor cortex, has been shown to negatively influence sensory acuity and motor control. The neuroplasticity underlying this reorganization may enhance the effectiveness of sensorimotor retraining therapies that involve specific stimulus features targeting somatosensory cortical regions.

This randomized controlled trial will include three groups: a device-assisted sensory acuity training group, a manual sensory acuity training group, and a control group receiving conventional physiotherapy. In this study, device-assisted sensory acuity training will be delivered using a standardized vibrotactile interface that presents controlled stimuli and records participant responses. The intervention will be structured to target sensory acuity components similar to those addressed in manual training.

Accordingly, the structured training protocol will include:

* localization training to improve detection of stimulus location,
* orientation discrimination to identify stimulus direction,
* temporal acuity training to distinguish timing differences between tactile stimuli and
* graphesthesia training to improve recognition of shapes or letters drawn on the skin through tactile input.

The primary aim of this study is to evaluate sensory acuity in individuals with CLBP and to determine the effects of a structured manual and technology-based sensory acuity training program, combined with conventional physiotherapy, on pain intensity (VAS), lumbar two-point discrimination, and a composite sensory acuity score.

We hypothesize that adding manual and technology-based structured sensory acuity training (SAT) program to a conventional physiotherapy regimen including motor control exercises will support central nervous system reorganization, improve sensory profiles, and lead to improvements in pain-related variables, disability, and quality of life.

Through this structured SAT program, we aim to provide an approach that evaluates and trains multiple dimensions of sensory acuity in CLBP, including localization, orientation, and temporal discrimination.

DETAILED DESCRIPTION:
This study consists of three research groups: the Technology-Based Sensory Acuity Training Group (T-SATG), the Manual Sensory Acuity Training Group (M-SATG), and the Control Group (CG). All groups will receive conventional physiotherapy for comparison purposes. In addition, a structured technological SAT program will be administered to the T-SATG, and a structured manual SAT program will be administered to the M-SATG, while the control group will receive a patient education (PE) program designed not to provide additional sensory stimulation. This approach will ensure equal session duration across all groups.

All individuals with non-specific chronic low back pain (NCLBP) will receive conventional physiotherapy for 30 minutes per day, three days a week, for four weeks. All patient admissions will be conducted under the guidance of the same physiotherapy team to ensure consistent implementation of the protocol and to maintain patient safety throughout the study. Participants will be asked to refrain from receiving any additional treatments for their lower back during the four-week intervention period, and any changes in medication type or dosage will be recorded.

In this study, the motor control exercise (MCE) program administered as part of conventional physiotherapy will aim to optimize control of the spine and pelvis through appropriate muscle activation, postural alignment, and movement integrity. The program is based on a graded progression system that emphasizes activation of the transversus abdominis and multifidus muscles. It will begin with fundamental exercises involving isolated contractions of these muscles, followed by more complex movements-such as bridging and quadruped exercises-that require coordinated activation of both muscles. During each session, the physiotherapist will guide participants to ensure correct exercise technique and provide necessary adjustments.

Individuals with non-specific chronic low back pain (CLBP) included in the T-SATG and M-SATG will receive sensory acuity training (SAT) for 30 minutes, three times per week, over a four-week period, with the difficulty level progressively increasing each week. This training program comprises four sensory acuity components delivered sequentially: Localization Acuity Training (LAT), Orientation Acuity Training (OAT), Temporal Acuity Training (TAT), and Graphesthesia Training (GT).

The sensory acuity training program will follow a structured weekly progression. During Weeks 1 and 2, participants will complete three core components of the training: Localization Acuity Training (LAT), Orientation Acuity Training (OAT), and Temporal Acuity Training (TAT). In Weeks 3 and 4, the same three components will continue, and Graphesthesia Training (GT) will be added to the protocol, expanding the program to four sensory acuity domains. This stepwise progression is designed to gradually increase training complexity and ensure the systematic development of sensory discrimination abilities across the four-week intervention period.

Localization Acuity Training (LAT) aims to improve the individual's ability to perceive applied stimuli and accurately identify their location. Orientation Acuity Training (OAT) focuses on enhancing the ability to distinguish the direction of two consecutive stimuli. Temporal Acuity Training (TAT) targets the ability to correctly determine the number of stimuli when two successive stimuli delivered to a single point differ in timing. Finally, Graphesthesia Training (GT) involves recognizing letters drawn on the skin and represents a complex process that requires not only tactile acuity but also cortical-level processing and mental representation of the letters.

For both groups, participants will be asked to visually mark their responses to the presented stimuli for each training parameter (LAT, OAT, TAT, GT). Participants in the T-SATG will indicate their responses through a tablet application synchronized with the device (TactiPain). The system will automatically record correct and incorrect responses. Participants in the M-SATG will be provided with a paper template containing designated areas representing the stimulus variables, and they will be instructed to mark the perceived stimulus features on this template. All responses will be collected by the physiotherapist at the end of each session and recorded. This procedure will ensure standardization of the response process and maintain measurement reliability in both training methods.

1. Technology-Assisted Sensory Acuity Training Group (T-SATG): The TactiPain device will be designed as a wearable waist belt containing 16 vibration motors (Pololu - Shaftless Mini Vibration Motor, 10 × 3.4 mm) placed between the last costa and the sacrum. The motors will be aligned in a 4 × 4 matrix according to the distances recommended in the literature. The combination of neoprene and cotton fabric will optimize both comfort and vibration transmission. The device will be integrated with a computer interface for the physiotherapist and a tablet application for the participant. The physiotherapist will be able to adjust the intensity of the vibration motors, the duration of each vibration, and the rest periods between vibrations during the session through the interface. The user screen will be simple and user-friendly, recording only the responses and response times. This innovative system, which offers a structured SAT protocol via vibration motors, aims to contribute scientifically to clinical decision-making processes by retraining sensory interaction mechanisms and reducing pain in individuals with NCLBP. During the training, vibration intensity will be adjusted to correspond to different maximum motor voltage levels. Vibration duration and inter-stimulus intervals will be progressively advanced from easier to more challenging levels based on participant performance. This structured progression is designed to allow the selection of parameters most appropriate to the individual's sensory perception profile and physiological responses, thereby optimizing the development of sensory acuity skills. Perceptual sensitivity to the vibrotactile stimuli and response accuracy will serve as the main progression criteria determining the continuation of training. This method is based on sensory training protocols recommended in the literature to enhance participants' stimulus identification and discrimination abilities.
2. Manual Sensory Acuity Training Group (M-SATG): During this training, the thin and thick tips of the Semmes-Weinstein monofilament will be used to vary stimulus intensity (pressure magnitude) and to provide two different stimulus levels in order to progressively increase difficulty. All SAT parameters (localization, orientation, temporal acuity, and graphesthesia) will be administered using sets generated randomly prior to each training session via the random.org program. This method is intended to prevent the development of habituation in participants. All responses will be recorded by the researcher to monitor weekly progress. During training, an adhesive grid template consisting of 16 holes will be placed on the participant's lumbar region between the last rib and the sacrum. A personalized adhesive grid template will be prepared for each participant, and the grid will be placed directly on the skin before each session.

ELIGIBILITY:
Inclusion Criteria:

* Age between 25-45 years
* No spinal fracture or acute disc herniation
* Pain duration ≥ 3 months
* Pain intensity ≥ 4/10
* Central Sensitization Scale (CSI) score ≥ 40
* No current psychiatric illness or cognitive impairment
* No contraindications to exercise

Exclusion Criteria:

* Serious spinal pathologies (lumbar stenosis, spondylolisthesis, tumor, infection, metastasis, osteoporotic fracture, severe structural deformities, inflammatory arthritis)
* Conditions with radicular involvement or neurological deficits (sciatica, nerve root compression)
* Systemic or neurological diseases (diabetes mellitus, neuromuscular diseases, serious central or peripheral nervous system diseases, epilepsy)
* Mental disorders
* Pregnancy
* Lower extremity injuries
* Spinal surgery within the last three years
* Chronic generalized pain syndromes (fibromyalgia, chronic fatigue syndrome)
* Individuals receiving other treatment for non-specific chronic low back pain during the study period.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2027-05-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Baseline (prior to the intervention), end of treatment (after the 12th session), and 6 months post-treatment.
  In order to evaluate the pain levels of the participants, the average pain intensity in the last 7 days will be evaluated with the Visual Analog Scale (VAS).
Two-Point Discrimination Test (TPDT) | Baseline (prior to the intervention), end of treatment (after the 12th session), and 6 months post-treatment.
  TPDT skill levels of individuals with CLI will be measured using a commercially available mechanical aesthesiometer (Baseline, 12-1480 Aesthesiometer).
Sensory Acuity Composite Score | Baseline (prior to the intervention), end of treatment (after the 12th session), and 6 months post-treatment.
  Localization, orientation, and temporal acuity accuracy (%) will be calculated by taking the average value of the sum of the levels. Evaluations will be made using the thick end of the monofilament. Each application will be performed in two sets of 20 repetitions in random order, each set including location, direction, and number of stimuli. Localization accuracy will be assessed using a locognosy test, which measures the percentage of correct responses by touching areas numbered 1 to 16 on a 4x4 grid, with participants pointing to the correct point on the figure.
Roland Morris Disability Questionnaire (RMDQ) | Baseline (prior to the intervention), end of treatment (after the 12th session), and 6 months post-treatment.
  The Roland Morris Disability Questionnaire (RMDQ), consisting of 24 questions focusing on regular activities of daily living, will be used to assess participants' disability levels. The total score ranges from 0 to 24, with higher scores reflecting increasing disability and scores exceeding 14 indicating severe disability.

SECONDARY OUTCOMES:
Pain Pressure Threshold (PPT) | Baseline (prior to the intervention), end of treatment (after the 12th session), and 6 months post-treatment.
  Pain pressure threshold level will be assessed using the Baseline® Dolorimeter - 22 pound Capacity, a digital algometer.
Left-Right Judgment Task (LRJT) | Baseline (prior to the intervention), end of treatment (after the 12th session), and 6 months post-treatment.
  In order to evaluate the participants' body awareness and laterality perception, the response time and accuracy rate regarding the direction of the images of the body will be measured with the Left-Right Judgment Task (LRJT) Recognise Online™ program.
Tampa Kinesiophobia Scale (TKS) | Baseline (prior to the intervention), end of treatment (after the 12th session), and 6 months post-treatment.
  The Tampa Kinesiophobia Scale (TKS) consisting of 17 questions including work-related activities, re-injury and fear-avoidance parameters will be used to assess participants' fear of movement. A score >37 indicates that the patient has symptoms of kinesiophobia.
Pain Catastrophizing Scale (PCS) | Baseline (prior to the intervention), end of treatment (after the 12th session), and 6 months post-treatment.
  The PCS will be used to assess participants' feelings and thoughts about pain and pain catastrophizing. If the cut-off value of the pain catastrophizing scale is equal to or greater than 17, the values are considered high, and if it is less than 17, it is considered low.
Joint Position Sense (JPS) | Baseline (prior to the intervention), end of treatment (after the 12th session), and 6 months post-treatment.
  All participants will have their full range of motion (ROM) measured using an inclinometer, with 50% of each movement set as the JPS evaluation target. The researcher will guide the participant from a neutral position to the target position (50% ROM) and ask them to hold this position for 5 seconds and memorize it. Then, they will return to the starting position, and the participant will be asked to actively return to the same target position. When the participant reaches the target, they will indicate this by saying "yes," and the JPS error will be calculated in degrees. Each test will be repeated three times, and the average value will be used.
Fremantle Back Awareness Questionnaire (FBAQ) | Baseline (prior to the intervention), end of treatment (after the 12th session), and 6 months post-treatment.
  Participants' awareness levels related to the waist area will be assessed with the Fremantle Back Awareness Questionnaire (FBAQ), which consists of 9 items. An increase in the score in the questionnaire indicates a decrease in awareness.
Central Sensitization Scale (CSS) | Baseline (prior to the intervention), end of treatment (after the 12th session), and 6 months post-treatment.
  Participants' clinical symptoms of central sensitization will be assessed with the Central Sensitization Scale (CSS), which consists of 25 items and is scored between 0 (never) and 4 (always). It has been shown that a score above 40 can detect the presence of central sensitization, and this score will also be used in the project inclusion criteria.
Short form-36 (SF-36) | Baseline (prior to the intervention), end of treatment (after the 12th session), and 6 months post-treatment.
  The 36 items are divided into 8 subscales and 2 composite domains. A weighted Likert scale is recommended for each subscale. Items in the subscales are summed to obtain a total score for each subscale or dimension. Each of the 8 total scores is linearly converted on a scale of 0 (negative health) to 100 (positive health) to provide a score for each subscale. Each subscale can be used independently. For each domain (physical and mental composite): Mean score = 50, Standard deviation = 10

CONTACTS AND LOCATIONS:
Overall Officials: AYSE GURLUK, PhD (c), Principal Investigator — Medipol University

IPD SHARING:
Plan to Share IPD: Undecided